CLINICAL TRIAL: NCT01362036
Title: Phase 1 Open-Label Dose-Escalating Study Evaluating the Safety and Preliminary Efficacy of TXA127 in Patients With Low/Intermediate-1 Risk Myelodysplastic Syndrome and Thrombocytopenia
Brief Title: Phase I Study Evaluating TXA127 in Low/Intermediate-1 Risk Myelodysplastic Syndrome and Thrombocytopenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment feasibility issues, new study in design
Sponsor: Tarix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXA127-2010-003
Record Dates: First submitted 2011-04-23; First posted 2011-05-27 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — angiotensin I (1-7)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TXA127 sc injectable (Experimental): All cohorts will recieve TXA127; Cohorts receive either 300, 600, or 900 ug/kg daily
  Interventions: Drug: TXA127

INTERVENTIONS:
Drug: TXA127 — Cohorts in this study will receive 300, 600, or 900 ug/kg daily by subcutaneous injection
  Other Names: Angiotensin 1-7

SUMMARY:
Phase 1, single-center, open-label, sequential cohort dose escalation study. This is a 3 + 3 design study involving at least 3 subjects in ascending dose cohorts, with subjects participating up to 10 weeks.

The overall study objectives are to evaluate the safety and tolerability of TXA127 in thrombocytopenic subjects with low or intermediate-1 risk MDS.

Evaluation of the platelet response and the erythroid and granulocytic responses to TXA127 will provide preliminary efficacy data.

DETAILED DESCRIPTION:
The hematopoietic properties demonstrated in the preclinical and clinical studies support the investigation of TXA127 to stimulate stem cell and progenitor cell proliferation. This is an exploratory study in a limited population of low or intermediate-1 MDS subjects who have platelet counts of ≤50 x 109/L to evaluate the effects of TXA127 on platelet response and on granulocytic and erythroid response.

Platelet response will be defined as complete and major as below:

* Complete platelet response: increase of platelet count to >100 x 109/L
* Major platelet response: increase of absolute platelet count by >30 x 109/L Other responses will be according to modified IWG MDS criteria (2006). Daily subcutaneous dosing of TXA will be carried out both in the clinic at scheduled visits and at home between clinic visits for a period fo 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS using the World Health Organization classification and Low or Intermediate-1 risk MDS using the IPSS
* The mean of two platelet counts taken during the 2-week Screening Period must be ≤50 x 109/L, with no individual non-transfused count >60 x 109/L. Platelet counts taken prior to Informed Consent may be used as one of the two counts taken within 2 weeks prior to study Day 1, but both counts must be obtained within 4 weeks of commencement of treatment.
* Subjects must be ≥18 years of age at the time of obtaining informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at the time of screening
* Adequate Liver Function, as evidenced by a serum bilirubin ≤2 times the laboratory upper limit of normal (ULN) (except for patients with a confirmed diagnosis of Gilbert's Disease), ALT and/or AST ≤3 times the laboratory ULN.
* A serum creatinine concentration ≤2 mg/dL

Exclusion Criteria:

* Currently receiving any treatment for MDS other than transfusions (last transfusion must be at least 4 weeks prior to treatment).
* If granulocyte and/or erythropoetic growth factors are currently being received, there should be a 4-week washout prior to treatment, and they may not be used during the study period.
* Concurrent active malignancy (other than controlled prostate cancer, in situ cervical cancer, or basal cell cancer of the skin)
* Prior history of bone marrow transplantation
* Unstable angina, uncontrolled congestive heart failure [NYHA > class II], uncontrolled hypertension [diastolic > 100 mmHg], uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction, or a QTc interval value >450ms.
* Received Anti-Thymocyte Globuline (ATG) within 6 months of screening
* Received hypomethylating agents, immunomodulating agents, histone deacetylase inhibitors, cyclosporine, or mycophenolate within 4 weeks of start of treatment
* Received IL-11 (oprelvekin) within 4 weeks before screening
* Have ever previously received rTPO, PEG-rHuMGDF, eltrombopag, or romiplostim
* Less than 4 weeks since receipt of any investigational agent (not FDA approved, for any indication)
* History of arterial thrombosis (e.g., stroke or transient ischemic attack) in the past year
* History of venous thrombosis that currently requires anti-coagulation therapy
* Female subjects who are pregnant or breastfeeding. Women of childbearing potential are required to have a positive HCG serum or urine pregnancy test performed 7 days prior to first study drug dose
* Women of childbearing potential who are unwilling to use an adequate form of contraception during the course of the study.
* Subjects with current alcohol abuse, illicit drug use, or any other condition (e.g., psychiatric disorder) that, in the opinion of the Investigator, may interfere with the patient's ability to comply with the study requirements or visit schedule.
* Subjects with a known sensitivity to any of the study medication components.
* Subjects known to have active HIV or known to be seropositive for HTLV-I.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (changes from baseline for safety parameters) of TXA127 in thrombocytopenic subjects with low or Intermediate-1 risk myelodysplastic syndrome (MDS). | Once or twice weekly during treatment and at follow-up visits. (up to 2 years)
  Evaluations performed during the study include vital signs and physical exam at all visits (twice/week for 4 weeks of treatment and at follow-up visits occurring 2 & 4 weeks following last treatment), blood chemistry, CBC, and platelet counts (once per week for 4 weeks, and at follow-up visits), concomitant medication and adverse event evaluations throughout the study period (8 weeks).
  Safety and tolerability will be assessed by incidence, severity, and changes from baseline of all relevant parameters including adverse events (AEs), laboratory values, and vital signs

SECONDARY OUTCOMES:
Evaluate the platelet response (change in platelet count from baseline) of thrombocytopenic subjects with low or intermediate-1 risk MDS receiving TXA127. | Twice Weekly during treatment and at follow-up visits (up to 2 years)
  Platelet counts and response will be evaluated twice per week at clinic visits during the treatment period (4 weeks), and again at the follow-up visits (week 6 and week 8).
Assess the erythroid and granulocytic response (change from baseline) to TXA127 in patients with low or intermediate-1 risk MDS. | Weekly during treatment and at follow-up visits (up to 2 years)
  Erythroid and granulocytic responses will be evaluated once weekly during the treatment period (first visit of each treatment week), and again at the follow-up clinic visits.

CONTACTS AND LOCATIONS:
Overall Officials: Gere S diZerega, MD, Study Chair — Sponsor - US Biotest Inc,
Locations (1):
- MD Anderson Leukemia Department, Houston, Texas, United States